CLINICAL TRIAL: NCT06548035
Title: Developing a Resiliency Intervention to Support Healthcare Workers Engaged in the Provision of HIV Care
Acronym: Qinisa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Wits Health Consortium (Pty) Ltd (Other)
Responsible Party: Principal Investigator, Christina Psaros, Associate Director, Behavioral Medicine Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024P001407; R34MH126753 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Stress; Burnout, Professional
Keywords: Nurses; HIV; Resiliency
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The control condition will be a one-time, ~90-minute, didactic stress management session (with no interventionist follow-up). The session will provide information on the four-component model of stress and the energy battery exercise (asks participants to reflect on stressors and things that offset stress).
- Intervention (Experimental): The intervention condition will consist of six one-hour group sessions. The sessions will provide information on topics including relaxation response, the components of stress, recuperative sleep, mindful awareness, resilience, and social support. Sessions will also include practice-based exercises (e.g., breathing exercises, mindfulness exercises). Participants will also have the option of accessing a closed WhatsApp group moderated by the interventionist. The interventionist will initiate chats in between group sessions to provide support to participants in practicing stress management skills. All intervention sessions will be delivered by a trained professional nurse, who will be trained and closely supervised by the study team members. Individual supervision will be provided at least bi-weekly, with opportunities for group supervision with US interventionists using the 3RP intervention in other studies as needed.
  Interventions: Behavioral: Adapted Relaxation Response Resiliency Program (3RP)

INTERVENTIONS:
Behavioral: Adapted Relaxation Response Resiliency Program (3RP) — The 3RP intervention is an integrated program of relaxation response (RR) eliciting meditation and mindfulness exercises, social support, cognitive skills training, and positive psychology focused on developing skills to reduce the stress response, elicit the relaxation response and enhance resiliency.
  Arms: Intervention

SUMMARY:
The purpose of this study is to pilot an adapted resiliency-based mind-body intervention (the Relaxation Response Resiliency Program; the 3RP) for nurses that care for people with HIV (PWH) in the public sector in South Africa (SA). In Phase 1 [NIH Grant Number: R34MH131426; Human Research Ethics Committee (HREC) Ethics Reference Number: 220813], the investigators conducted focus group discussions to solicit feedback on: the role of culture and perceptions of stress; the lived experiences of stress; sources of stress (e.g. occupational, trauma related); how stress impacts job functioning (specifically patient care); current coping strategies; and the intervention modules (content, number of sessions, session duration, program length, mode of delivery (e.g., virtual, in-person, hybrid approaches, use of coaches), etc.). In this phase 2, the investigators will conduct a small proof-of-concept study (N = 8-10), followed by a randomized pilot (N = 60) of nurses that care for PWH in the public sector in South Africa (SA) to test the feasibility and acceptability of the adapted intervention.

DETAILED DESCRIPTION:
This study will pilot test an adapted version of an existing stress management and resiliency-enhancing intervention (the Relaxation Response Resiliency Program; the 3RP) for nurses that care for PWH in the public sector in SA, to test the feasibility and acceptability of all study procedures. This intervention was adapted and refined from its original format (which consisted of eight, 90-minute weekly group sessions) following focus group discussions (FGDs) that explored nurses' preferences and desired modifications to the intervention (Phase 1 of this study).

This trial will involve a randomized pilot study (N = 60) to test the feasibility and acceptability of the adapted intervention among nurses that care for PWH in the public sector in SA.

Additionally, the randomized control trial (RCT) will collect anonymous clinic client data on demographics, satisfaction with care, client-provider trust, and likelihood of returning to care. We will also collect clinic-level data to understand how to measure client-related outcomes and clinic metrics of HIV care engagement, such as expected patient return rates/measures of retention, percentage of patients with suppressed viral load, frequency of viral load collection, and percentage of patients initiating second line treatment to best understand how to measure these variables in a larger trial testing the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Providing at least some primary HIV care in a public sector clinic (at the level of professional nurse) for at least one year;
* IsiZulu or English speaking;
* Able and willing to sign informed consent.

Exclusion Criteria:

- Participation in cognitive behavioral therapy and/or a mind-body intervention in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of Study Procedures, as Assessed by Number of Individuals Enrolled and Number of Assessments and Sessions Completed by Enrolled Individuals. | Through study completion, approximately 12 months after initiation
  To assess feasibility, the investigators will track the number of participants screened, eligible, and enrolled; the number of treatment and assessment sessions completed; and reasons for declining enrollment and for prematurely leaving the trial.
Acceptability of Study Procedures, as Assessed by the Client Satisfaction Questionnaire | Immediately after the intervention
  Acceptability will be measured through the Client Satisfaction Questionnaire (CSQ-8): 8-item measure of how much one values an intervention. Items scored from 1 (poor) to 4 (excellent); higher scores indicate greater satisfaction. Totals range from 8 to 32; with scores between 26 and 32 indicating 'excellent acceptability' and scores between 20 and 25 indicating 'good acceptability'. High internal consistency (alpha = 0.84-0.93) and used in HIV intervention research and resource-limited settings.
Acceptability of Study Procedures | Immediately after the intervention
  Acceptability will also be assessed via qualitative exit interviews.

SECONDARY OUTCOMES:
Resilience | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Measure of Current Status (MOCS-A): 13-item measure of stress reactivity and coping; statements are rated from 0 (I cannot do this at all) to 4 (I can do this extremely well); total score ranges from 0-52; higher scores suggest better coping skills. Current Experiences Scale (CES): 25-item measure of resiliency domains; scores range from 0-125; higher scores reflect greater resilience.
Perceived Stress | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Perceived Stress Scale (PSS-10): 10-item measure of the extent to which past month life situations are appraised as stressful. Scores range from 0-40; higher scores indicate higher perceived stress.
Burnout | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Maslach Burnout Inventory Human Services Survey for Medical Personnel (MBI-HSS [MP]): 22-item measure of job burnout in medical professionals. The MBI-HSS comprised 22 questions across 3 subscales; Emotional Exhaustion (EE)-9 questions, Depersonalization (DP)-5 questions, and self-perceived lack of Personal Accomplishment (PA)-8 questions.
  High scores on the emotional exhaustion and depersonalization dimensions correspond to higher levels of burnout and high scores on the personal accomplishment dimension refer to lower levels of burnout.
Absenteeism | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention.
  Absenteeism will be measured by assessing unplanned days off from work in the prior 30 days.
Compassion Fatigue | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Professional Quality of Life Scale (ProQOL) Version 5: 20-item burnout and secondary traumatic stress subscales from larger 30-item measure. Subscale scores range from 10-50; higher scores represent greater burnout and secondary traumatic stress.
Stigma | Baseline
  Measuring HIV Stigma and Discrimination Among Health Facility Staff: Standardized Brief Questionnaire (BL). Higher score represent greater stigma.
Anxiety | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Generalized Anxiety Disorder (GAD-7) scale: 7- item measure of the severity of anxiety symptoms over the past two weeks. Scores range from 0-21; cutoff scores of 5, 10, and 15 indicate mild, moderate, and severe anxiety.
Depression | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Patient Health Questionnaire (PHQ-9): 9-item tool to evaluate the presence and frequency of depressive symptoms in the past two weeks. Scores range from 0-27; cutoffs of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depression.
Social Support | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Coping Orientation to Problems Experienced (COPE) Inventory: Two 4-item subscales of the 53-item COPE Inventory (use of emotional support, use of instrumental support) to assess frequency of use of social support to cope with stress. Subscale scores range from 4-16, with higher scores indicating greater use of emotional or instrumental support.
Optimism | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Life Orientation Test - Revised (LOT-R): 10-item measure of generalized optimism vs. pessimism about the future. Total scores range from 0-24; higher scores indicate greater optimism.
Distress Tolerance | Baseline, pre-intervention; immediately after the intervention; 3 months after the intervention
  Distress Tolerance Scale (DTS): 15-item measure. Total scores range from 15-75; higher scores indicate greater distress tolerance.
  of emotional distress tolerance.
Adherence to 3RP intervention skills | Weeks 1-6 of intervention
  Practice notes have been developed to correspond with each module of the 3RP treatment.
  Participants will be asked to keep brief daily diaries of their out-of-session practice of core skills, which will be used to generate a rating of adherence to out-of-session practice guidelines. Note, completion will be encouraged but is not required.

CONTACTS AND LOCATIONS:
Locations (1):
- MatCh Research nit (MRU), a Division of Wits Health Consort, Durban, South Africa

IPD SHARING:
Plan to Share IPD: No